CLINICAL TRIAL: NCT01315717
Title: Maladie d'Alzheimer et Troubles Locomoteurs : Caracterisation Des Anomalies Temporelles de la Marche et Etude Des Correlats Anatomo-cognitifs
Brief Title: Gait and Alzheimer Interaction Tracking (GAIT) Study
Acronym: GAIT
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2009-A00533-54
Record Dates: First submitted 2011-03-10; First posted 2011-03-15 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2011-03

CONDITIONS: Gait Apraxia; Alzheimer Disease; Impaired Cognition; Cerebral Atrophy
MeSH Terms: conditions — Gait Apraxia; Alzheimer Disease; Cognition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group 1: Healthy subjects
- Group 2: Patients with Mild Cognitive Impairment
- Group 3: Patients with Mild AD
- Group 4: Patients with Moderate AD

SUMMARY:
The purpose of this study is to examine and to compare gait characteristics under single- and dual-task conditions among healthy subjects together with AD patients at different stages of disease (i.e., pre-dementia, mild and moderate dementia stages).

DETAILED DESCRIPTION:
Although gait disorders are frequently associated with Alzheimer's disease (AD), few studies have focused on their characterization and mechanism. Exploring the associations of the gait characteristics - more particularly the gait variability - with the cognitive performance of AD patients on one hand, and with the morphological brain abnormalities on the other hand, could be useful to understanding the mechanisms of gait disorders in AD.

The main objective of this study is to examine and to compare gait characteristics under single- and dual-task conditions among healthy subjects together with AD patients at different stages of disease (i.e., pre-dementia, mild and moderate dementia stages).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Able to walk without walking aid on 15 metres
* Score of Mini-Mental Examination (MMSE) > 10
* Written informed consent to participate in the study (or trustworthy person)
* Being affiliated to a social security regime
* Near visual acuity ≥ 2/10
* Absence of severe depression (score in the 15-item Geriatric Depression Scale ≤ 10)

Exclusion Criteria:

* Score of Mini-Mental Examination (MMSE) ≤ 10
* Subject suffering from pre-existing impellent disturbances
* History of cerebrovascular accident or other cerebro-spinal pathology
* Poor workmanship of the written or oral French language
* Refusal of subject to be informed on possible hanging bare anomaly during study
* Use of walking aid
* Acute medical or surgical disease in the past 3 months
* Refusal to participate (or trustworthy person)
* Contra-indication to the achievement of a Magnetic Resonance Imaging
* Near visual acuity < 2/10
* Presence of severe depression (score in the 15-item Geriatric Depression Scale > 10)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients of the University Memory Center of Angers Hospital with respect to the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 912 (Actual)
Dates: Start 2009-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Stride-to-stride variability of stride time | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, PhD, Principal Investigator — Angers University Hospital
Locations (1):
- Angers University Hospital, Angers, France

REFERENCES:
- [Derived] Graffe A, Beauchet O, Fantino B, Milea D, Annweiler C. Vitamin D and macular thickness in the elderly: an optical coherence tomography study. Invest Ophthalmol Vis Sci. 2014 Jul 15;55(8):5298-303. doi: 10.1167/iovs.14-13918. PMID 25028353